CLINICAL TRIAL: NCT03116581
Title: Study on the Parameters That Influence Perceptual Decisions
Brief Title: Altruistic Decisions
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient on-site staff to manage study
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL16_0680
Record Dates: First submitted 2017-03-07; First posted 2017-04-17 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Healthy
Keywords: Perceptual Decision; Social Cognition; Motivation
MeSH Terms: interventions — Magnetoencephalography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vicarious reward (Other): If a decision influences the well-being of another (through monetary payoff), the decision making processes should differ from a decision that would influences only oneself. The difference will be reflected in the reaction-times and in the accuracy of the response to the task. The drift diffusion models care then used to estimate le decision parameter in each condition and understand which parameter is influenced by the beneficiary of the payoff associated with a decision.
  Once the decision parameter characterized with behavioral experiment, the study aims to better understand the neural network sustaining the influence of others on the decision making process, by assessing the neural activity related to the decision making processes. Also, the research compares how the brain responses for payoff for others and payoffs for oneself, specially to confirm that these responses are located in different areas of the Anterior cingulate Cortex.
  Interventions: Other: Behavior; Other: fMRI (functional Magnetic Resonance Imagery); Other: MEG (MagnetoEncephaloGraphy)
- Audience effect (Other): In order to clarify the complex changes in the decision-making processes induced by simple observation by others (audience) , the experiment have two levels of difficulty . These levels of difficulty will be determined in such a way as to achieve better 'public' performance than 'private' when the task is easy (high level of consistency) and poor performance when the task is difficult (low level of coherence) As described in the literature in psychology. Drift diffusion models will be used to better understand the variations in performance, to decipher between a modulation of the diffusion velocity and or of the decision threshold. This study will help characterize how observation by others modulates performance. Once the decision parameter characterized with behavioral experiment, the study aims to better understand the neural network sustaining the impact of observation by others on the decision making process.
  Interventions: Other: Behavior; Other: fMRI (functional Magnetic Resonance Imagery); Other: MEG (MagnetoEncephaloGraphy)

INTERVENTIONS:
Other: Behavior — Random-dots tasks: dots appear and move, most have a random trajectory but a given proportion of them move coherently to the same direction.
  * Vicarious reward Each trial begins with a cue, showing 'me' or 'him' and filled rectangle filled proportionally to the payoff. The cue and the square are depicted in yellow (oneself) or blue (other), depending on the beneficiary. The moving dots are then presented and the subjects respond. At the end of dots motion, the feedback is presented. If the response was correct, a pile of coins proportional to the payoff is shown. For incorrect responses and misses, a red-colored cross is displayed.
  * Audience effect Each trial begins with the display of two eyes (public) or a padlock (private). The moving dots are shown and the participant answers. Audience condition changes the information available on accuracy when submitting comments. In the observed condition, an arrow shows the response. In the observed condition, no feedback is displayed.
Other: fMRI (functional Magnetic Resonance Imagery) — Both behavioral task (audience effect and vicarious reward) will be studied in fMRI (functional Magnetic Resonance Imagery). The same paradigms used in the behavioral experiment will be adapted for fMRI.
  Audience Effect experiment: trials will last for 10 seconds maximum. With 80 trials for each condition (public easy, public difficult, private easy and private difficult), the task will count a total of 320 trials and have a 54 minutes duration, in 3 runs of 17 minutes each.
  Vicarious Reward experiment: trials will have a 10 seconds maximum duration. Using 40 trials for each condition (other low payoff, other high payoff, self low payoff, self high payoff, control condition), the task will have a total of 200 trials and last for 54 minutes, in 6 runs of 9 minutes each.
Other: MEG (MagnetoEncephaloGraphy) — Both behavioral task (audience effect and vicarious reward) will be studied in MEG (MagnetoEncephaloGraphy). The same paradigms used in the behavioral experiment will be used in MEG.
  Audience Effect experiment: trials will last for 7 seconds maximum. With 100 trials for each condition (public easy, public difficult, private easy and private difficult), the task will count a total of 400 trials and have a 47 minutes duration. Every 100 trials (about 12 minutes of tasks), a break will be proposed to the participants.
  Vicarious Reward experiment: trials will have a 7.2 seconds maximum duration. Using 75 trials for each condition (other low payoff, other high payoff, self low payoff, self high payoff, control condition), the task will have a total of 375 trials and last for 45 minutes. Every 125 trials (every 15 minutes), a break will be proposed to the participants.

SUMMARY:
The study aimed to understand how payoffs for others influence perceptual decision making. The research consists in testing how varying monetary payoffs for another modify the perceptual decision making processes. The use of drift diffusion models on a random dots task enable the characterization of the decision parameter(s) that are modulated when a decision is made to win payoffs for others as compared to decisions for self-benefits. Once the parameter revealed through behavioral experiment, neuroimaging is applied to find the neural correlates of the effects of taking others into account in the decision making process.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 35
* Right-handed
* French
* Normal vision or corrected by contact lenses

Exclusion Criteria:

* Contraindications to the MEG examination
* Presence of a perceptual disorder (vision) or motor impairing the capacity to carry out the tasks requested (including dyschromatopsia and achromatopsia).
* Taking of medical treatment in progress (excluding contraceptive pill).
* Known neurological or psychiatric history or disorders.
* Participants in an exclusion period for any other research.
* Participants who do not benefit from social protection.
* Participants refusing to be informed of the results of the medical examination.
* Participants who refuse to be informed of the possible detection of an anomaly.
* Participants with MRI contraindications

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 159 (Actual)
Dates: Start 2014-02-03 (Actual); Primary Completion 2016-07-22 (Actual); Study Completion 2016-07-22 (Actual)

PRIMARY OUTCOMES:
Modulation of the decisional parameter by the payoff conditions | 1 hour
  behavioral data (reaction-times and accuracy) are collected and the decision parameter can be estimated from them using Drift Diffusion Models
Modulation of the decisional parameter by the beneficiary conditions | 1 hour
  behavioral data (reaction-times and accuracy) are collected and the decision parameter can be estimated from them using Drift Diffusion Models

SECONDARY OUTCOMES:
Event-Related potentials | 1 hour
  study of the time-locked brain activity
Time-frequency brain responses | 1 hour
  study of the oscillatory activity elicited in the brain
BOLD | 1 hour
  Variation of the blood-oxygen-level dependent (BOLD) signal

CONTACTS AND LOCATIONS:
Overall Officials: Caroline DEMILY, MD, Principal Investigator — CH le Vinatier
Locations (1):
- CH le Vinatier, Bron, France